CLINICAL TRIAL: NCT06525350
Title: A Randomized, Controlled, Open-label Phase Ⅱ Study to Evaluate the Safety, Tolerability, and Efficacy of the Combination of Glumetinib Tablets and Docetaxel for Injection（Albumin Bound）Verse Docetaxel in the Treatment of Locally Advanced/Recurrent or Distant Metastasized Non-small Cell Lung Cancer Patients With MET Overexpression
Brief Title: A Study to Evaluate the Efficacy and Safety of the Combination of Glumetinib and Docetaxel（Albumin Bound）Verse Docetaxel for the Treatment of MET-overexpressed Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SYH2065-001
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced/Recurrent or Distant Metastasized Non-small Cell Lung Cancer With MET Overexpression
MeSH Terms: conditions — Recurrence | interventions — glumetinib; Docetaxel

STUDY DESIGN:
Intervention Model Description: In stage 2, participants who meet the eligibility criteria are randomly assigned to the experimental group (glumetinib tablets+HB1801), factorial group (glumetinib tablets), and control group (docetaxel) in a 2:1:1 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glumetinib tablets+HB1801 combination treatment arm (Experimental): Glumetinib tablets RP2D PO QD, HB1801 RP2D iv Q3W until a treatment discontinuation criterion is met.
  Interventions: Drug: Glumetinib tablets; Drug: HB1801 (docetaxel, albumin-bound）
- Glumetinib tablets monotherapy arm (Experimental): Glumetinib tablets RP2D PO QD until a treatment discontinuation criterion is met.
  Interventions: Drug: Glumetinib tablets
- Docetaxel monotherapy arm (Active Comparator): Docetaxel 75mg/m^2 iv Q3W until a treatment discontinuation criterion is met.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Glumetinib tablets — An ATP competitive, highly selective MET receptor tyrosine kinase inhibitor
  Arms: Glumetinib tablets monotherapy arm; Glumetinib tablets+HB1801 combination treatment arm
Drug: HB1801 (docetaxel, albumin-bound） — An improved new formulations of docetaxel
  Arms: Glumetinib tablets+HB1801 combination treatment arm
Drug: Docetaxel — A chemotherapy drug
  Arms: Docetaxel monotherapy arm

SUMMARY:
This study consists of Stage 1 (including dose escalation and dose expansion) and Stage 2 (randomized controlled study). The main purpose of Stage 1 is to preliminarily evaluate the safety and tolerability of the combination of glumetinib Tablets and Docetaxel for Injection（Albumin Bound）(HB1801) in the treatment of MET-overexpressed non-small cell lung cancer (NSCLC); The main purpose of Stage 2 is to evaluate the efficacy of the combination of glumetinib tablets and HB1801 compared to glumetinib tablets monotherapy or docetaxel in the treatment of MET-expressed NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and voluntarily sign a written informed consent form;
* 2. Age ≥ 18 years old, gender unlimited;
* 3. Unresectable locally advanced or metastatic non-small cell lung cancer (IIIB, IIIC, or IV according to the 8th edition TNM staging standards of IASLC) confirmed by histology or cytology;
* 4. Participants must provide tumor tissue samples that meet the testing requirements of the central laboratory, or agree to accept the tumor tissue biopsy, used for central laboratory testing of MET expression and amplification, and the development of MET associated diagnostic reagents;
* 5. Confirmation of MET overexpression in tumor tissue specimens through the central laboratory designated by the sponsor;
* 6. Driver genes alterations must be negative (including EGFR mutations, ALK fusion, ROS1 rearrangement fusion, BRAF V600 mutation, NTRK fusion, MET 14 exon skipping mutation, RET rearrangement, HER2 Mutations, KRAS activation mutations, etc.);
* 7. Previously received immunotherapy with PD-1/PD-L1 monoclonal antibody and platinum-containing chemotherapy (combination therapy or sequential therapy);
* 8. At least one measurable lesion exists at the baseline that meets the definition of RECIST 1.1;
* 9. ECOG performance score of 0 or 1;
* 10.Expected survival time ≥ 3 months;
* 11.Adequate organs and bone marrow function within 7 days prior to initial administration.

Exclusion Criteria:

* 1. Previously received MET-targeted drug therapy;
* 2. Previous treatments included docetaxel;
* 3. Existence of meningeal metastasis, spinal cord compression, or active and untreated brain metastasis;
* 4. Imaging evidence of clear tumor cavity, capsule or large vessel invasion, and tumor adjacent to important vascular structures , Which has been determined by researchers that there is a risk of fatal bleeding;
* 5. Suffering from central squamous cell lung cancer with cavities or hemoptysis (>50 mL/d);
* 6. Within 14 days before the first administration, there is an uncontrollable accumulation of serous cavity effusion that requires frequent drainage or medical intervention;
* 7. Adverse reactions from previous anti-tumor treatments (including radiotherapy) have not yet recovered to ≤ level 1(according to CTCAE 5.0) or baseline level (excluding toxicity assessed by researchers as having no safety risk such as hair loss, fatigue, pigmentation, etc);
* 8. Suffering from other malignant tumors within 5 years prior to the first administration. (Except already treated local tumors, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ and breast carcinoma in situ);
* 9. Received any systemic anti-tumor therapy within 28 days or 5 half-lives prior to initial administration (whichever is shorter) treatment, including chemotherapy, targeted therapy, biological therapy, immunotherapy, immunomodulatory drugs (including thymosin, interleukin-2, interferon, tumor necrosis factor, etc.), or other research drugs;
* 10. Received radiation therapy involving the chest cavity within 28 days prior to the first administration, o received radiation therapy not involving the chest cavity within 14 days prior to the first administration;
* 11. Received Chinese herbal medicine or traditional Chinese patent medicines for tumor control within 14 days before the first administration;
* 12. Received potent cytochrome P450 3A4 (CYP3A4) inhibitor or induction within 14 days prior to initial administration or Patients who cannot suspend the use of CYP3A4 potent inhibitors during the study;
* 13. Having undergone major surgery (excluding biopsy) or severe traumatic damage within 28 days before the first administration, or expected to undergo major surgery during the study;
* 14. A history of gastrointestinal perforation and/or fistula, severe gastrointestinal ulcers or surgery, gastrointestinal dysfunction, or other diseases that may affect the absorption of experimental drugs within 6 months prior to the first administration;
* 15. Existence of ≥ grade 2 edema and lymphedema that cannot be relieved through clinical intervention;
* 16. Received live vaccine or attenuated live vaccine within 28 days prior to initial administration or planned to receive live vaccine or attenuated live vaccine during the study period;
* 17. Within 14 days prior to the first administration, there is a need of systemic antibiotics, antifungal or antiviral for the treatment of severe chronic or active infections (including tuberculosis infections, etc.);
* 18. Severe or uncontrollable cardiovascular diseases that require treatment 6 months before screening;
* 19. Interstitial lung disease (ILD) or drug-induced interstitial pneumonia, non-infectious pneumonia, including radiation pneumonia, pulmonary fibrosis, or acute lung disease that require steroid treatment;
* 20. History of immunodeficiency, including human immunodeficiency virus (HIV) infection or known acquired immunodeficiency history of AIDS, or other acquired or congenital immunodeficiency diseases, or organ transplantation history;
* 21. Active hepatitis B, active hepatitis C, active syphilis or active Tuberculosis;
* 22. History of autoimmune diseases;
* 23. Previous serious illnesses;
* 24.Known to have allergies or hypersensitivity reactions to any investigational drug or any investigational drug excipients, or other serious allergy history;
* 25. Breastfeeding or pregnant women; The blood pregnancy test conducted by women with fertility within 7 days prior to enrollment in the trial is positive;
* 26. Any male and female patients with fertility who refuse to use highly effective contraceptive methods during the entire trial period and 6 months after the last administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) occurrence and incidence | Up to approximately 48 months after the first participant is enrolled
Recommended phase 2 dose(RP2D) of the combination therapy | Up to approximately 48 months after the first participant is enrolled
Adverse events (AE) and serious adverse events (SAE) occurrence and incidence | Up to approximately 48 months after the first participant is enrolled
Objective response rate (ORR) per RECIST 1.1 | Up to approximately 48 months after the first participant is enrolled

SECONDARY OUTCOMES:
Disease control rate (DCR) per RECIST 1.1 | Up to approximately 48 months after the first participant is enrolled
Duration of response (DoR) per RECIST 1.1 | Up to approximately 48 months after the first participant is enrolled
Progression free survival (PFS) per RECIST 1.1 | Up to approximately 48 months after the first participant is enrolled
Blood drug concentrations of glumetinib and HB1801 | Up to approximately 48 months after the first participant is enrolled
MET expression level | Up to approximately 48 months after the first participant is enrolled
MET amplification level | Up to approximately 48 months after the first participant is enrolled
Tumor-associated gene variations | Up to approximately 48 months after the first participant is enrolled
Overall survival(OS) | Up to approximately 48 months after the first participant is enrolled